CLINICAL TRIAL: NCT00866320
Title: A Phase II Study of Sorafenib in Patients With Metastatic Renal Cell Carcinoma (RCC) Refractory to SU11248 or Bevacizumab Therapy
Brief Title: Sorafenib in Treating Patients With Metastatic Kidney Cancer That Has Not Responded to Sunitinib or Bevacizumab
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE11805; P30CA043703 (NIH); CASE11805 (Other: Case Comprehensive Cancer Center); 05-167 (Other: Cleveland Clinic IRB)
Record Dates: First submitted 2009-03-19; First posted 2009-03-20 (Estimated); Results first posted 2012-02-01 (Estimated); Last update posted 2014-07-23 (Estimated); Status verified 2014-07

CONDITIONS: Kidney Cancer
Keywords: clear cell renal cell carcinoma; recurrent renal cell cancer; stage IV renal cell cancer
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sorafenib (Experimental): Chemotherapy single agent systemic. Sorafenib given up to 600mg orally every 12 hours for up to 10 months (40 weeks).
  Interventions: Drug: sorafenib tosylate

INTERVENTIONS:
Drug: sorafenib tosylate — Sorafenib (BAY 43-9006) is an oral multi-kinase inhibitor targeting both tumor cells and the tumor vasculature. Patients with metastatic RCC meeting eligibility criteria will receive 400 mg BID of sorafenib in a single-arm phase II study. Treatment will be administered on an outpatient basis.

SUMMARY:
RATIONALE: Sorafenib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor.

PURPOSE: This phase II trial is studying how well sorafenib works in treating patients with metastatic kidney cancer that has not responded to sunitinib or bevacizumab.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the tumor burden reduction rate in patients with sunitinib malate- or bevacizumab-refractory, metastatic clear cell renal cell carcinoma treated with sorafenib tosylate.

Secondary

* To determine the safety of sorafenib tosylate in these patients.
* To record the duration of tumor reduction, time to disease progression, and overall survival of patients treated with sorafenib tosylate.

OUTLINE: Patients receive oral sorafenib tosylate twice daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed renal cell carcinoma with a component of clear cell histology

  * Metastatic disease
* Disease progression, as defined by RECIST criteria, after prior treatment with sunitinib malate or bevacizumab

  * Patients must have received ≥ 1 course (4 weeks) of sunitinib malate or ≥ 2 doses of bevacizumab AND have RECIST-defined objective progression during or within 4 months after completing treatment with sunitinib malate or bevacizumab
* Measurable disease by RECIST criteria
* CNS metastases allowed provided patient has undergone prior surgery and/or radiotherapy AND has no evidence of further CNS disease progression by CT scan or MRI ≥ 2 weeks after treatment of CNS metastases

PATIENT CHARACTERISTICS:

* ECOG performance status (PS) 0-1 or Karnofsky PS 70-100%
* WBC ≥ 3,000/μL
* Absolute neutrophil count ≥ 1,500/μL
* Platelet count ≥ 75,000/μL
* Total bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST/ALT ≤ 2.5 times ULN
* Creatinine ≤ 2.0 times ULN
* Negative pregnancy test
* No significant cardiovascular disease, including any of the following:

  * Congestive heart failure (New York Heart Association class III-IV heart disease)
  * Active angina pectoris requiring nitrate therapy
  * Uncontrolled dysrhythmias
  * Cardiovascular event within the past 6 months (e.g., transient ischemic attack/cerebrovascular accident, myocardial infarction, or vascular surgery)

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* At least 2 weeks since prior systemic therapy, radiotherapy, or major surgery and recovered
* No prior sorafenib tosylate
* No other concurrent investigational agents
* No other concurrent anticancer therapy
* No concurrent prophylactic growth factors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2006-02; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian I. Rini, MD, Principal Investigator — Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center
Locations (2):
- United States (2):
  - Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio
  - Baylor Sammons Cancer Center, Dallas, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is a multiple site study. Patients were recruited 2/2006-4/2008 from medical hospitals in Cleveland, Ohio and Dallas, Texas
Groups:
- Sorafenib: Patients receive Sorafenib 400 mg BID until disease progression or toxicity. Dose may be escalated to 600mg and 800 mg BID after the 8 week disease reassessment.
Period: Overall Study
Arm/Group | Sorafenib
Started | 49
Completed | 43 (All patients that received treatment were analyzed.)
Not Completed | 6
Not completed — Withdrawal by Subject | 4
Not completed — Death | 2

BASELINE CHARACTERISTICS:
Arm/Group | Sorafenib
Number analyzed (Participants) | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.2 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 13
Region of Enrollment [Number; unit: participants]
  United States | 49

OUTCOME MEASURES:

1. Primary Outcome: Tumor Burden Reduction Rate (TBRR)
Description: The primary endpoint of the study is defined as the percentage of patients who experience larger than or equal to 5% reduction in tumor burden as measured by RECIST-defined target lesions without progression of non-target lesions or the appearance of any new lesions, confirmed at least 4 weeks after first documentation. RECIST criteria will be used for the purpose of designating target lesions, calculating total tumor burden (the sum of the unidimensional measurement of target lesions) and defining disease progression.Additional RECIST-defined partial or complete responses will be recorded.
Time Frame: at 8 weeks (2cycles of treatment)
Population: All patients who started treatment
Measure: Number; unit: percentage of patients
Groups:
- Sorafenib: Patients receive sorafenib twice a day until disease progression or toxicity.
Arm/Group | Sorafenib
Number analyzed (Participants) | 47
percentage of patients
  Achieved at least 5% tumor reduction | 30
  Did not achieve at least 5% tumor reduction | 70

2. Secondary Outcome: Overall Survival
Description: Overall survival measured in months and summarized using the Kaplan-Meier method. This will be calculated from the date of registration on-study to the dates of documented evidence of progression and death, respectively.
Time Frame: followed until progression or death for approximately 3 years
Population: All patients who started treatment
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sorafenib
Number analyzed (Participants) | 47
months | 16 [7.6 to 32.3]

3. Secondary Outcome: Time to Progression
Description: Time to objective progression will be measured from the start of treatment until the criteria for RECIST-defined progression are met, taking as reference the smallest measurements recorded since the treatment started, including baseline.
  Progression-free survival measured in months and summarized using the Kaplan-Meier method.
Time Frame: followed to progression for approximately 3 years
Population: All patients who started treatment
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Sorafenib: Sorafenib twice a day until progression or toxicity
Arm/Group | Sorafenib
Number analyzed (Participants) | 47
months | 4.4 [3.6 to 5.9]

4. Secondary Outcome: Duration of Overall Response (Tumor Burden Reduction)
Description: Measured from the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented.
Time Frame: followed for overall response for approximately 3 years
Population: Patients who achieved at least 5% tumor reduction
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sorafenib
Number analyzed (Participants) | 14
months | 7.1 [2.1 to 9.2]

ADVERSE EVENTS:
Time Frame: Adverse events collected from the start of treatment to the end of the study for a period of 3 years and 8 months.
Arm/Group | Sorafenib
Serious Adverse Events (participants affected / at risk) | 4/47
Other Adverse Events (participants affected / at risk) | 41/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sorafenib (N=47)
Anorexia (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Constitutional Symptoms (General disorders) | 1
Hand-Foot Skin Reaction (Skin and subcutaneous tissue disorders) | 1
Metabolic/Laboratory (Metabolism and nutrition disorders) | 1
Myalgia (muscle pain) (Musculoskeletal and connective tissue disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Pain (General disorders) | 1
Thrombosis/embolism (Cardiac disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sorafenib (N=47)
Hemoglobin (Blood and lymphatic system disorders) | 4
Hypertension (Vascular disorders) | 16
Edema (General disorders) | 4
Fatigue (General disorders) | 25 — Lethargy, malaise, asthenia
Fever (General disorders) | 3 — Fever (in the absence of neutropenia, where neutropenia is defined as AGC<1.0 x 10e9/L)
Rigors, Chills (General disorders) | 3
Weight Loss (General disorders) | 10
Alopecia (Skin and subcutaneous tissue disorders) | 12
Rash/desquamation (Skin and subcutaneous tissue disorders) | 14
Dry Skin (Skin and subcutaneous tissue disorders) | 6
Hand-Foot Skin Reaction (Skin and subcutaneous tissue disorders) | 28
Dermatology/Skin-other (Skin and subcutaneous tissue disorders) | 14
Hypothyroidism (Endocrine disorders) | 4
Anorexia (Gastrointestinal disorders) | 17
Constipation (Gastrointestinal disorders) | 5
Diarrhea (Gastrointestinal disorders) | 25 — patients without colostomy
Taste Disturbance (dysgeusia) (Gastrointestinal disorders) | 7
Nausea (Gastrointestinal disorders) | 13
Stomatitis/pharyngitis (Gastrointestinal disorders) | 13 — oral/pharyngeal mucositis
Vomiting (Gastrointestinal disorders) | 6
Gastrointestinal-other (Gastrointestinal disorders) | 11
General Disorders-other (General disorders) | 3
Musculoskeletal-other (Musculoskeletal and connective tissue disorders) | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 — Joint pain
Headache (Nervous system disorders) | 4
Myalgia (muscle pain) (Musculoskeletal and connective tissue disorders) | 5
Pain-other (General disorders) | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 — shortness of breath
Voice Changes/stridor/larynx (Reproductive system and breast disorders) | 4 — hoarseness, loss of voice, laryngitis

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes